CLINICAL TRIAL: NCT06784895
Title: Designing and Assessing a Women Only Cardiac Rehabilitation Program
Brief Title: Designing and Assessing a Women Only Cardiac Rehabilitation (CARE) Program
Acronym: CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Texas (Other)
Responsible Party: Principal Investigator, Melvyn Rubenfire, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00252649
Record Dates: First submitted 2025-01-16; First posted 2025-01-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Rehabilitation; Cardiovascular Diseases
Keywords: Female only CR program; Standard of care rehab program; Education sessions
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study team will make every effort to:
  * Mask the Cardiopulmonary Exercise Test (CPET)/Volume of Oxygen consumed (VO2) test technicians that will be administering these assessments from knowing which treatment arm the participant is receiving.
  * Mask the registered dietician as to which study participants are in the control group and are receiving the standard CR programming (unable to blind for experimental group due to the nature of the group CR sessions)
  * Mask the statistician as to which group received which CR programming during data analysis.
  * Limit contact and conversation between participants and non-CR staff; example lab technicians, nurses, medical assistants, and dietitians
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women only Cardiac Rehab program (Experimental)
  Interventions: Behavioral: Women only Cardiac Rehab program
- Standard of Care (mixed-sex) rehab program (Active Comparator)
  Interventions: Behavioral: Standard of Care (mixed-sex) rehab program

INTERVENTIONS:
Behavioral: Women only Cardiac Rehab program — This is a 12-week program and will include 36 sessions 3 times a week. This group will also have Women-Only Education sessions. Participants will also have a 24-week follow-up visit from the time of entry.
  Women-specific education content will be provided monthly in addition to the standard weekly "mini-teaches." This education content will be developed and delivered by experience health care professionals that are experts in women's health.
  Arms: Women only Cardiac Rehab program
Behavioral: Standard of Care (mixed-sex) rehab program — This is a 12-week program and will include up to 36 sessions 3 times a week. Participants will also have a 24-week follow-up visit from the time of entry. Exercise classes are medically supervised, and each program is individualized based upon medical history, cardiac risk factors, goals, and initial fitness level. Educational programs are arranged in a continuing series, with sessions taught by experts in nutrition therapy, stress reduction therapy, and exercise.
  Arms: Standard of Care (mixed-sex) rehab program

SUMMARY:
The purpose of this randomized controlled study is to investigate the effect(s) of a pilot women-only cardiac rehabilitation (CR) program. The study team will be testing the effectiveness, compliance and enjoyment of this women's only cardiac rehabilitation (CR) program by comparing outcomes to those randomized to receive Michigan Medicine's current CR program (standard care), which includes people of all genders.

Study hypotheses:

* Women randomized to women-specific CR programming will have superior attendance and completion rates compared to women attending mixed-sex CR programming.
* Women randomized to women-specific CR programming will experience greater improvement in clinical outcomes in comparison to those in mixed-sex CR programming.

DETAILED DESCRIPTION:
This registration was updated on 11/24/2025 due to amendments that were approved at the IRBMED.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability to participate in study procedures for the duration of the study
* Identify as a female
* Be between the ages of 40-80 years, inclusive
* Documented diagnosis of CR indications of stable angina pectoris, acute myocardial infarction (MI) within the preceding 6 months, percutaneous coronary interventions (PCI), surgical and transvalvular aortic valve replacement, post-aortic surgery with or without aortic valve, coronary artery bypass grafting (CABG) and mitral valve replacement or repair with or without CABG
* Referred to outpatient CR at the University of Michigan, Domino's Farms or Brighton Center for Specialty Care Cardiac Rehabilitation site based on Michigan Medicine's Division of Cardiovascular Medicine Policy and Procedure.

Exclusion Criteria:

* Not being "cleared" for CR based on Michigan Medicine's Division of Cardiovascular Medicine Policy and Procedures
* Prior participation in CR
* Inability to understand spoken and written English, either due to language barrier or cognitive limitation for any reason, including deaf or blind
* Frailty, fall risk, or muscle, joint or back pain as defined as the inability to perform activities of daily living without limitations and engage in mild physical activity (i.e. unable to walk up 1 flight of stairs unaided)
* Any of the following as the indication for CR: aortic repair or replacement for aortic dissection, untreated or greater than New York Heart Association (NYHA) class II congestive heart failure, coronary artery dissection without coronary artery disease, fibromuscular hyperplasia, stress cardiomyopathy, cardiac transplant candidate or recipient
* Life threatening ventricular arrythmias without an implanted defibrillator; very frequent premature ventricular contraction or premature atrial contractions symptomatic or not; poorly controlled atrial fibrillation
* Associated more than mild valvular heart disease, untreated congestive heart failure; unstable angina or heart pain with minimal activity; angina or congestive heart failure limiting ability to climb one flight of stairs without help (NHYA Functional Classification >2)
* Severe pulmonary hypertension (right heart systolic pressure greater than 60 millimeters of mercury); clot in the heart; treated venous thrombosis with or without pulmonary embolism in past 6 months; more than mild dyspnea related to chronic lung disease or asthma
* Chronic kidney disease (creatinine >2 milligrams per deciliter (mg/dl)); symptomatic active liver disease (infectious or inflammatory), symptomatic chronic liver disease (except for nonalcoholic fatty liver disease), kidney dialysis or kidney transplant recipient, active or chronic renal disease (rise by 0.5mg/dL in past 3 months or chronic elevated serum creatinine 2.0 milligrams per milliliter (mg/mL) or greater.
* Poorly controlled diabetes defined as uninterrupted HbA1c >8.0% for ≥1 year despite standard care, baseline HbA1c prior to CR > 8.5%.
* Immunosuppressive drug requirement, acute anemia, chronic anemia with Hemoglobin < 10mg/mL
* Limiting chronic muscle, joint, or back pain; identified as fall risk from poor balance or neurologic syndromes; frailty defined as the inability to perform activities of daily living in older adults that carries an increased risk for poor health outcomes including falls, incident disability, hospitalization, and mortality
* Untreated or active substance abuse/addiction including alcohol and drugs; depression (defined as a score ≥ 15 or depression positive answer to #8 or #9 on Patient Health Questionnaire-9) unless deemed acceptable by mental health care provider; severe anxiety
* Severe obesity (Body mass index ≥ 40 kilograms/meters squared), on weight loss drugs (unless target body weight has been achieved or use is for glycemic control in diabetes), history of bariatric surgery; chronic venous insufficiency with cellulitis or > 1+ edema unless controlled with support hose.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cardiac Rehabilitation (CR) attendance rate | 12 weeks (post CR)
  CR completion rate defined as number of patients that "graduated" or completed CR programming versus the number of patients that started CR programming [i.e. attended 75% or more of the prescribed sessions (≥27 out of 36)], expressed as a percentage of participants per arm.
Cardiac Rehabilitation (CR) attendance rate - percentage | 12 weeks (post CR)
  Number of CR sessions attended out of number of CR sessions prescribed, expressed as a percentage

SECONDARY OUTCOMES:
Optimal blood pressure (BP) control | 12 weeks (post CR)
  Percentage of patients that have optimal BP control at program discharge, defined as systolic blood pressure (SBP) less than 130 mmHg and diastolic blood pressure (DBP) less than 80 Millimeters of mercury (mmHg).
Change in resting systolic blood pressure (SBP) | Baseline, 12 weeks (post CR)
  Change in resting SBP from baseline to CR completion, measured using an automated blood pressure monitor and expressed in mmHg.
Change in resting diastolic blood pressure (DBP) | Baseline, 12 weeks (post CR)
  Change in resting DBP from baseline to CR completion, measured using an automated blood pressure monitor and expressed in mmHg.
Improvement in depression based on the Patient Health Questionnaire (PHQ)-9 | Baseline to 12 weeks (post CR)
  Percentage (%) of patients with a positive depressive screen at CR entrance that experience a decrease in depressive symptoms (reduction in one or more levels of severity) as measured by changes in the Patient Health Questionnaire (PHQ)-9 score from baseline to completion of CR.
  The PHQ-9 questionnaire is a self-assessed questionnaire that asks participants to respond to 9 questions with response options of 0, 1, 2 or 3. The total score scale ranges from 0 to 27. Higher scores indicate more symptoms of depression.
Change in Patient Health Questionnaire (PHQ)-9 score | Baseline to 12 weeks (post CR)
  A change in PHQ-9 scores will be measured during the first 12 weeks of the study. The PHQ-9 questionnaire is a self-assessed questionnaire that asks participants to respond to 9 questions with response options of 0, 1, 2 or 3. The total score scale ranges from 0 to 27. Higher scores indicate more symptoms of depression.
Change in Patient Health Questionnaire (PHQ)-9 score | 12 weeks (post CR), 24 weeks
  The PHQ-9 questionnaire is a self-assessed questionnaire that asks participants to respond to 9 questions with response options of 0, 1, 2 or 3. The total score scale ranges from 0 to 27. Higher scores indicate more symptoms of depression. A change in PHQ-9 scores will be measured during the first 12 weeks of the study and will be repeated 12 weeks following program completion.
Improvement in functional capacity measured by the six-minute walk test | Baseline, up to 12 weeks (post CR)
  Percentage of patients that achieve an increase in distance walked, in meters, by at least 10%, after participation in CR as measured by the 6-minute walk test (6MWT).
Change in 6-minute walk test distance | Baseline, 12 weeks (post CR)
  The distance walked in six minutes on a standard course will be measured in meters at baseline and CR Exit
Improvement in functional capacity Metabolic Equivalents (METs) | Baseline, 12 weeks (post CR)
  Percentage of patients that display an overall mean increase in estimated METs (0.93 METs, 12.4%): with greatest increase occurring in "low" fitness patients < 5 METs (1.3 METs, 35% increase), followed by "moderate" fitness 5-8 METs (1.03 METs, 16% increase), and "high" fitness > 8 METs (0.77 METs, 8% increase)2,3 after participation in CR as measured by estimated exercise session peak METs.
Change in estimated exercise session peak METs | Baseline, up to 12 weeks (post CR)
  The difference in estimated peak METs between baseline (defined as the third session to account for learning effect) and program completion.

CONTACTS AND LOCATIONS:
Overall Officials: Melvyn Rubenfire, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No